CLINICAL TRIAL: NCT06186167
Title: Histopathological Incidence of Amyloidosis in High-Risk Patients Undergoing Cardiac Device Implantation
Brief Title: Amyloidosis Incidence in High-Risk Cardiac Device Patients
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Midwest Heart & Vascular Specialists (Other)
Responsible Party: Sponsor
Other Study IDs: MWHV-AMYLO-BIOP-001
Record Dates: First submitted 2023-12-16; First posted 2023-12-29 (Actual); Last update posted 2024-02-20 (Actual); Status verified 2023-12

CONDITIONS: Amyloid; Cardiac Amyloidosis; Amyloidosis Cardiac; Systemic Amyloidosis; AL Amyloidosis; Infiltrative Cardiomyopathy, Amyloid; ATTR Amyloidosis Wild Type
Keywords: Cardiac Devices; Chest Wall Fat Pad Biopsy; Cardiac Implantable Electronic Devices
MeSH Terms: conditions — Alzheimer Disease; Amyloid Neuropathies, Familial; Immunoglobulin Light-chain Amyloidosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — The biospecimens consist of chest wall fat tissue samples collected during cardiac device implantation procedures. This adipose tissue, typically excised to create space for the device, is preserved for histopathological analysis to detect amyloid deposits. The analysis of these samples is crucial for diagnosing cardiac amyloidosis in patients at high risk. The tissue will be handled and analyzed by the HCA pathology laboratory, following standard procedures to ensure the integrity of the samples and the accuracy of the diagnostic results.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

GROUPS / COHORTS (1):
- High-Risk Cardiac Device Recipients: Participants in this cohort are individuals undergoing clinically indicated cardiac device implantation, such as pacemakers, ICDs, ILRs, or CRT-D/Ps. During the standard implantation procedure, chest wall fat tissue typically excised to create space for the device is collected for histopathological analysis to identify amyloid deposits. This study involves no additional intervention beyond the routine clinical care received by the patients.
  Interventions: Procedure: Chest Wall Fat Tissue Collection

INTERVENTIONS:
Procedure: Chest Wall Fat Tissue Collection — As part of routine cardiac device implantation, chest wall fat tissue is collected for histopathological analysis. This tissue, which is typically discarded, will be used to identify amyloid deposits in high-risk cardiac patients. No additional surgical intervention is performed beyond the standard procedure for device implantation.

SUMMARY:
This single-practice prospective cohort study aims to enhance the diagnosis of cardiac amyloidosis in high-risk patients undergoing standard cardiac device implantation. By analyzing chest wall fat tissue, which is usually discarded, we aim to determine the diagnostic yield of such biopsies for amyloidosis and to develop a predictive screening model based on clinical, lab, and imaging data. The study, running from December 2023 to December 2024, expects to enroll 100 patients and may provide a new, non-invasive diagnostic avenue for this condition.

DETAILED DESCRIPTION:
The study targets a key gap in cardiac amyloidosis diagnosis by systematically evaluating the histopathological incidence of the disease using chest wall fat pad biopsies-tissue that is typically discarded during the implantation of cardiac devices like pacemakers, ICDs, and CRT-D/Ps. Standard surgical procedures are adhered to, ensuring minimal additional risk to patients. The collected tissue samples are analyzed by the HCA pathology laboratory to detect amyloid deposits, thereby potentially identifying amyloidosis in a non-invasive manner. In addition to the primary endpoint of histopathological diagnosis, the study retrospectively aims to validate a predictive model that incorporates a wide range of data to streamline the identification of patients at high risk for cardiac amyloidosis. Strict measures are in place to protect patient confidentiality and data security. By potentially improving diagnostic efficiency, this research could contribute to earlier detection and treatment strategies, thus improving patient outcomes for those at high risk of this life-threatening condition.

ELIGIBILITY:
Inclusion Criteria:

* Patients who are 40 years of age or older
* Patients who are able and willing to provide informed consent
* Patients who are scheduled for CIED implantation within the study period and with clinical lab and imaging features suggestive of cardiac amyloidosis

Exclusion Criteria:

* Individuals below the age of 40.
* Persons who are unable to consent or who do not consent to participate.
* Patients who have already been diagnosed with cardiac amyloidosis prior to the study

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: High-risk patients undergoing cardiac device implantation who meet the study's inclusion criteria.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2024-01-29 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Diagnostic yield of chest wall fat pad biopsy for cardiac amyloidosis | December 2023 to December 2024, corresponding to the study duration during which patients will be enrolled and outcomes will be assessed
  The primary outcome measure is the histopathologic diagnosis of amyloidosis in chest wall fat tissue removed during cardiac device implantation

SECONDARY OUTCOMES:
Development of a predictive screening model for cardiac amyloidosis | Retrospective analysis of patient data collected from December 2023 to December 2024
  Retrospective development and validation of a predictive model using pre-procedural clinical, lab, and imaging data to identify patients at high risk for cardiac amyloidosis

CONTACTS AND LOCATIONS:
Overall Officials: Vasvi Singh, MD, Principal Investigator — Midwest Heart & Vascular Specialists
Locations (1):
- Midwest Heart & Vascular Specialists, Overland Park, Kansas, United States

IPD SHARING:
Plan to Share IPD: Undecided
At present, the specifics of a data-sharing plan for individual participant data (IPD) from this study are under consideration. The study team intends to protect patient confidentiality and data integrity and will comply with all relevant regulations and guidelines for data sharing. Once a plan has been established, details about the nature of the data to be shared, the conditions for access, and the timing for data release will be provided.

REFERENCES:
- [Background] Takano R, Ueda N, Okada A, Matsumoto M, Ikeda Y, Hatakeyama K, Izumi C, Kusano K. Fat biopsy from a pocket of cardiac implantable electronic device: An alternative diagnostic option for cardiac amyloidosis. HeartRhythm Case Rep. 2022 May 18;8(8):554-557. doi: 10.1016/j.hrcr.2022.05.008. eCollection 2022 Aug. No abstract available. PMID 35996711